CLINICAL TRIAL: NCT01937858
Title: The Correlation Between HbA1c and Mean Blood Glucose in Patients With Diabetes and Renal Failure
Status: Terminated | Type: Observational
Sponsor: Reem Mohammad Alamoudi (Other)
Responsible Party: Sponsor-Investigator, Reem Mohammad Alamoudi, Consultant Endocrinology, King Abdullah International Medical Research Center
Organization: King Abdullah International Medical Research Center (Other)
Other Study IDs: RC08/107/A
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Diabetes; Renal Failure
Keywords: HbA1c; glycated hemoglobin; correlation; diabetes; renal failure
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal renal function
- Stage 2 and 4 and 5 chronic kidney disease
- End stage renal disease on hemodialysis

SUMMARY:
The value of HbA1c as a tool to determine glycemic control in patients with diabetes and renal failure has not been well studied, the same accepted normal ranges for HbA1c are applied to all patients with diabetes regardless of their renal function. We would like to evaluate the use of HbA1c as a tool of assessing long term glycemic control in this subgroup of patients with diabetes and evaluate the effect of dialysis on HbA1c

ELIGIBILITY:
Inclusion Criteria:

All patients >18 years of age with type 1 or 2 diabetes who show competence in home glucose monitoring and are willing to commit to doing the testing

Exclusion Criteria:

* Pregnancy
* Having received a blood transfusion with in the preceding three months
* Known to have any hereditary or hemolytic anemia
* On a medication known to interfere with HbA1c assay (opiates, acetaminophen, vitamin C, vitamin E) - we will allow patients to be on asprin as almost all patients with diabetes are on this drug.
* Having a blood hemoglobin <7 mg/dl
* Bilirubin level >20mg/dL or a triglyceride level > 250mg/dL
* Alcohol addiction

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our target population is patients with diabetes and impaired renal function. This study will include 80 adult patients with type1 or type 2 diabetes; 20 with normal serum creatinine, 40 with renal failure in the predialysis stage (20 with stage 3 and 4 CKD [GFR 0f 20-40] and 20 with stage 5 CKD not yet on hemodialysis [GFR <20]), and 20 on hemodialysis. All patients should be comfortable and committed to doing self-glucose monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Correlation | three months
  The quantitative correlation between mean blood glucose and HbA1c in patients with diabetes and renal failure